CLINICAL TRIAL: NCT04995926
Title: Efficiency and Safety of Labial Mucosal Epithelium Grafting for Corneal Reepithelization in Patients With Bilateral Non-immunogenic Limbal Stem Cell Deficiency
Brief Title: Labial Mucosal Epithelium Grafting for Corneal Limbus Substitution
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The S.N. Fyodorov Eye Microsurgery State Institution (Other Government)
Responsible Party: Principal Investigator, Boris Malyugin, Deputy Director of Science, The S.N. Fyodorov Eye Microsurgery State Institution
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 517062021
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Limbal Stem-cell Deficiency
Keywords: Limbal Stem Cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Labial mucosa epithelium grafting for corneal limbus substitution. (Experimental): Surgery for treating limbal stem cell deficiency using a strip of the lip oral mucosa with trimmed off the substantia propria and grafted as a circular corneal limbus substitute.
  Interventions: Procedure: Labial mucosal epithelium grafting for corneal limbus substitution

INTERVENTIONS:
Procedure: Labial mucosal epithelium grafting for corneal limbus substitution — Labial mucosa epithelium grafting for corneal limbus substitution will be used to treat limbal stem cell deficiency by way of corneal surface re-epithelization

SUMMARY:
Earlier approaches for cornea reepithelization in patients with bilateral LSCD included allogeneic corneal limbus grafting from postmortem donor or livingrelated relatives with concomitant systemic immunosuppression (Cheung and Holland, 2017) and cultivated oral mucosal epithelial transplantation (COMET) (Nishida et al., 2004).

The novel surgical technique for corneal re-epithelization were described by Liu et al. (2011) and Choe et al. (2019). In both clinical studies, the autologous labial mucosal epithelium graft was transplanted as a surrogate corneal limbus for purpose of treatment the LSCD. Authors reported positive outcomes in terms of anatomical success and corneal status improvement.

The purpose of the study is to evaluate the feasibility of the novel surgical intervention in clinical use.

DETAILED DESCRIPTION:
Earlier approaches for cornea reepithelization in patients with bilateral LSCD included allogeneic corneal limbus grafting from postmortem donor or livingrelated relatives with concomitant systemic immunosuppression (Cheung and Holland, 2017) and cultivated oral mucosal epithelial transplantation (COMET) (Nishida et al., 2004).

The novel surgical technique for corneal re-epithelization were described by Liu et al. (2011) and Choe et al. (2019). In both clinical studies, the autologous labial mucosal epithelium graft was transplanted as a surrogate corneal limbus for purpose of treatment the LSCD. Authors reported positive outcomes in terms of anatomical success and corneal status improvement.

Lip oral mucosa is a promising autologous source of epithelial cell for the trial because it has similar histological characteristic as the normal corneal. In particular, lip oral mucosal epithelium is stratified squamous and nonkeratinized.

The indicated histological and molecular features of the lip oral mucosal epithelium predetermined the use of labial mucosal epithelial graft for treatment patients with bilateral LSCD.

The purpose of the study is to confirm the validity of the hypothesis about the possibility of re-epithelialization diseased cornea using labial mucosal epithelium graft as a surrogate limbus in patients with bilateral LSCD.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman 18 years and older.
* Signed informed consent, given by the participant or his/her legal representative.
* Ability to understand Russian spoken and written language.
* Sanitated oral cavity.
* Bilateral limbal stem cell deficiency diagnosed by two or more symptoms during slit-lamp examination: corneal conjunctivalization, absence of palisades of Vogt, superficial corneal neovascularization, recurrent or persistent corneal epithelium erosion.
* Bilateral limbal stem cell deficiency non-immunogenic etiology (burns, irradiation, contact lens related, etc.).
* Best-corrected visual acuity less than 0.3 (6/18 Snellen chart)
* Intraocular pressure in normal range.
* Schirmer's test I more than 5 mm.

Exclusion Criteria:

* Inability to give signed informed consent.
* Age under 18 years.
* Pregnancy and/or breastfeeding.
* Hormonal contraceptives intake.
* History of allergic reactions to antibiotics, glucocorticosteroids, remedies for treatment dry eye syndrome, medications for local and general anesthesia.
* Participation in other clinical trials.
* Systemic immunosuppression intake.
* Diagnosed neoplastic process or treatment for it.
* Positive tests for infectious: HIV, syphilis, Hepatitis B, Hepatitis C.
* Any medical, psychiatric and/or condition, including cachexia, or social conditions that the investigator believes would interfere with or contraindicate adherence to the research protocol or the ability to provide signed informed consent.
* Immune-mediated limbal stem cell deficiency (Stevens-Johnson syndrome, ocular cicatricial pemphigoid and other.), unknown and/or inherited etiology.
* Best-corrected visual acuity more than 0.3 (6/18 Snellen chart)
* Ocular burns earlier than 12 months.
* Keratoplasty earlier than 12 months.
* Limbal grafting (from postmortem or living-related donors).
* Keratoprosthetic device or history of its implantation.
* Cellular therapy for treatment of limbal stem cell deficiency.
* Cellular transplantation for treatment of limbal stem cell deficiency.
* Active ophthalmic infection.
* Symblepharon, ectropion, trichiasis, lagophthalmos and/or other lid and/or conjunctival fornixes abnormalities.
* Surgery on ocular adnexa earlier than 9 months.
* Corneal stromal thickness less than 300 mkm.
* Dry eye with Schirmer test I less than 5 mm and/or keratinized ocular surface.
* Uncontrolled glaucoma and/or presents of a glaucoma drainage device.
* Retinal defunctioning (no light perception and/or retinal detachment).
* Absence of the electric activity of the optic nerve and/or retina.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Anatomical success | 12 months
  Presence of a stable epithelium on the cornea and absence of conjunctivalization in the visual axis of the recipient eye

SECONDARY OUTCOMES:
Number of participants with improvement in corneal status | 12 months
  A composite score for the corneal disease status (Campbell et. al., 2019) of the patients will be obtained throughout the study using the following 4 criteria in points according to the grades (grade 0, grade 1 - mild, grade 2 - moderate, grade 3 - severe):
  1. corneal staining: 0 - no punctuate staining, 1 - superficial punctate keratopathy (SPK) less than 50% of the corneal surface, 2 - SPK more than 50% of the corneal surface, 3 - epithelial defect;
  2. conjunctivalisation: 0 - absent, 1 - <25% of corneal surface, 2 - 25-50% of corneal surface, 3 - >50% of corneal surface;
  3. corneal neovascularization: 0 - absent, 1 - confined to corneal periphery, 2 - extending to pupil margin, 3 - extending beyond pupil margin into central cornea;
  4. corneal opacification: 0 - clear cornea, iris details clearly visualized, 1 - partial obscuration of iris details, 2 - iris details poorly seen with pupil margin just visible, 3 - complete obscuration of iris and pupil details.
Functional success | 12 months
  Improvement in near and/or distance visual acuity
Rate of complications | 12 months
  Intraoperative and postoperative complications on the recipient eye

CONTACTS AND LOCATIONS:
Overall Officials: Boris E Malyugin, MD PhD Prof, Principal Investigator — The S. Fyodorov Eye Microsurgery Federal State Institution
Locations (1):
- The S. Fyodorov Eye Microsurgery Federal State Institution, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
We plan to share Clinical Study Report, present and publish results of the study.
Supporting Information: CSR
Time Frame: During the study and after.
Access Criteria: upon request

REFERENCES:
- [Background] Malyugin B.E., Borzenok S.A., Gerasimov M.Y. Clinical outcomes of autologous cultured oral mucosal epithelium transplantation for treatment of limbal stem cell deficiency. Fyodorov Journal of Ophthalmic Surgery. 2020;(4):77-85. (In Russ.) doi:10.25276/0235-4160-2020-4-77-85
- [Background] Borzenok S.A., Gerasimov M.Yu., Ostrovskiy D.S., Malyugin B.E. Culture of human labial mucosal epithelial cell for use in patients with bilateral limbal stem cell deficiency. Russian Journal of Transplantology and Artificial Organs. 2019;21(3):111-120. doi:10.15825/1995-1191-2019-3-111-120
- [Background] Cabral JV, Jackson CJ, Utheim TP, Jirsova K. Ex vivo cultivated oral mucosal epithelial cell transplantation for limbal stem cell deficiency: a review. Stem Cell Res Ther. 2020 Jul 21;11(1):301. doi: 10.1186/s13287-020-01783-8. PMID 32693830
- [Background] Campbell JDM, Ahmad S, Agrawal A, Bienek C, Atkinson A, Mcgowan NWA, Kaye S, Mantry S, Ramaesh K, Glover A, Pelly J, MacRury C, MacDonald M, Hargreaves E, Barry J, Drain J, Cuthbertson B, Nerurkar L, Downing I, Fraser AR, Turner ML, Dhillon B. Allogeneic Ex Vivo Expanded Corneal Epithelial Stem Cell Transplantation: A Randomized Controlled Clinical Trial. Stem Cells Transl Med. 2019 Apr;8(4):323-331. doi: 10.1002/sctm.18-0140. Epub 2019 Jan 28. PMID 30688407
- [Background] Choe HR, Yoon CH, Kim MK. Ocular Surface Reconstruction Using Circumferentially-trephined Autologous Oral Mucosal Graft Transplantation in Limbal Stem Cell Deficiency. Korean J Ophthalmol. 2019 Feb;33(1):16-25. doi: 10.3341/kjo.2018.0111. PMID 30746908
- [Background] Deng SX, Borderie V, Chan CC, Dana R, Figueiredo FC, Gomes JAP, Pellegrini G, Shimmura S, Kruse FE; and The International Limbal Stem Cell Deficiency Working Group. Global Consensus on Definition, Classification, Diagnosis, and Staging of Limbal Stem Cell Deficiency. Cornea. 2019 Mar;38(3):364-375. doi: 10.1097/ICO.0000000000001820. PMID 30614902
- [Background] Deng SX, Kruse F, Gomes JAP, Chan CC, Daya S, Dana R, Figueiredo FC, Kinoshita S, Rama P, Sangwan V, Slomovic AR, Tan D; and the International Limbal Stem Cell Deficiency Working Group. Global Consensus on the Management of Limbal Stem Cell Deficiency. Cornea. 2020 Oct;39(10):1291-1302. doi: 10.1097/ICO.0000000000002358. PMID 32639314
- [Background] Holland EJ, Mogilishetty G, Skeens HM, Hair DB, Neff KD, Biber JM, Chan CC. Systemic immunosuppression in ocular surface stem cell transplantation: results of a 10-year experience. Cornea. 2012 Jun;31(6):655-61. doi: 10.1097/ICO.0b013e31823f8b0c. PMID 22333664
- [Background] Inamochi A, Tomioka A, Kitamoto K, Miyai T, Usui T, Aihara M, Yamagami S. Simple oral mucosal epithelial transplantation in a rabbit model. Sci Rep. 2019 Dec 2;9(1):18088. doi: 10.1038/s41598-019-54571-7. PMID 31792300
- [Background] Li W, Li Q, Wang W, Li K, Ling S, Yang Y, Liang L. A rat model of autologous oral mucosal epithelial transplantation for corneal limbal stem cell failure. Eye Sci. 2014 Mar;29(1):1-5. PMID 26016058
- [Background] Liu J, Sheha H, Fu Y, Giegengack M, Tseng SC. Oral mucosal graft with amniotic membrane transplantation for total limbal stem cell deficiency. Am J Ophthalmol. 2011 Nov;152(5):739-47.e1. doi: 10.1016/j.ajo.2011.03.037. Epub 2011 Jul 30. PMID 21803325
- [Background] Nakamura T, Endo K, Cooper LJ, Fullwood NJ, Tanifuji N, Tsuzuki M, Koizumi N, Inatomi T, Sano Y, Kinoshita S. The successful culture and autologous transplantation of rabbit oral mucosal epithelial cells on amniotic membrane. Invest Ophthalmol Vis Sci. 2003 Jan;44(1):106-16. doi: 10.1167/iovs.02-0195. PMID 12506062
- [Background] Nishida K, Yamato M, Hayashida Y, Watanabe K, Yamamoto K, Adachi E, Nagai S, Kikuchi A, Maeda N, Watanabe H, Okano T, Tano Y. Corneal reconstruction with tissue-engineered cell sheets composed of autologous oral mucosal epithelium. N Engl J Med. 2004 Sep 16;351(12):1187-96. doi: 10.1056/NEJMoa040455. PMID 15371576
- [Background] Oliva J, Bardag-Gorce F, Niihara Y. Clinical Trials of Limbal Stem Cell Deficiency Treated with Oral Mucosal Epithelial Cells. Int J Mol Sci. 2020 Jan 9;21(2):411. doi: 10.3390/ijms21020411. PMID 31936462